CLINICAL TRIAL: NCT03323502
Title: A Nursing Home Pragmatic Trial of APPROACHES (Aligning Patient Preferences: a Role Offering Alzheimer's Patients, Caregivers, and Healthcare Providers Educ. and Support)
Brief Title: Aligning Patient Preferences: a Role Offering Alzheimer's Patients, Caregivers, and Healthcare Providers Education and Support
Acronym: APPROACHES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: National Institute on Aging (NIA) (NIH); Hebrew SeniorLife (Other); Regenstrief Institute, Inc. (Other)
Responsible Party: Principal Investigator, Susan Elizabeth Hickman, Professor, Community Health Systems, Indiana University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 00481769; R21AG057463-01 (NIH)
Record Dates: First submitted 2017-10-24; First posted 2017-10-27 (Actual); Results first posted 2025-08-26 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-11

CONDITIONS: Alzheimer Disease; Dementia
Keywords: Nursing Homes; Skilled Nursing Facilities; Advance Care Planning; Advance Directives; Alzheimer Disease; Dementia; Do Not Resuscitate Orders; Physician Orders for Life-Sustaining Treatment; Artificial Nutrition; Hospitalization; Intubation; Pragmatic Clinical Trials; Randomized Controlled Trials; Patient Preferences; Resuscitation Orders
MeSH Terms: conditions — Alzheimer Disease; Dementia; Patient Preference | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: Behavioral: ACP Specialist Program
Masking Description: Cluster Randomized Pragmatic Trial: Randomization will occur at the facility level. In order to implement the intervention in the treatment arms facilities, study staff will be required to know the identity of participating facilities. Since this trial involves training staff at intervention facilities, the masking will be 'open label'.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- APPROACHES ACP Specialist Program (Experimental): Enrolled facilities that will be trained in the APPROACHES Advance Care Planning (ACP) Specialist Program.
  Interventions: Behavioral: APPROACHES ACP Specialist Program
- Control (Active Comparator): Enrolled facilities that will perform standard of care Advance Care Planning (ACP) procedures.
  Interventions: Other: Standard of care

INTERVENTIONS:
Behavioral: APPROACHES ACP Specialist Program — The APPROACHES Advance Care Planning (ACP) Specialist will work with nursing home leaders (in intervention arm facilities) to: i. Consolidate nursing home ACP procedures; ii. Train and educate staff; and iii. Facilitate ACP Specialist Program with patients who have Alzheimer's disease/related dementias and their family caregivers.
  Arms: APPROACHES ACP Specialist Program
Other: Standard of care — Standard of care Advance Care Planning (ACP) procedures
  Arms: Control

SUMMARY:
Nursing home (NH) patients with Alzheimer's disease and related dementias often receive unwanted, burdensome treatments such as hospitalization. Advance care planning (ACP) is a key strategy to support patients and family-caregivers in making informed decisions and ensuring treatment preferences are proactively known and honored. The ACP Specialist Program will improve care and reduce unwanted, burdensome hospitalizations through improved ACP procedures, standardized staff education on ACP, and systematic ACP facilitation delivered by existing NH staff.

DETAILED DESCRIPTION:
A significant number of patients with Alzheimer's disease or related dementia diagnoses will be cared for in nursing homes near the end of life. Unfortunately, many of these patients experience unwanted and burdensome medical treatments, such as potentially avoidable hospitalizations, that negatively impact quality of life. Advance care planning (ACP) discussions with patients and family caregivers are important to explore goals in advance of a crisis and support informed, values-based decision-making. The ACP process helps ensure that preferences about treatments such as hospitalization are known, documented, and honored. Research indicates that ACP can reduce burdensome treatments and increase the likelihood that care will match documented preferences. Nursing homes are currently required by regulations to offer ACP to patients and families. However, there are no training requirements for nursing home staff and approaches to fulfilling this regulatory and ethical responsibility vary widely, resulting in inconsistent ACP. The "Aligning Patient Preferences - a Role Offering Alzheimer's patients, Caregivers, and Healthcare providers Education and Support (APPROACHES)" trial will test the APPROACHES ACP Specialist Program. Existing nursing home staff members will be trained to enhance care and reduce unwanted, burdensome hospitalizations through improved ACP procedures, standardized staff education on ACP, and systematic ACP facilitation. The primary trial outcome is annual hospital transfers (admissions and emergency department visits). Consistent with the spirit of a pragmatic trial, study outcomes rely on data already collected for quality improvement, clinical or billing purposes. In the 18 month R21 pilot phase, the aims are to: 1) Establish the trial's organizational structure and processes; and 2) Pilot test the intervention in 4 nursing homes. In the R33 phase, a pragmatic cluster randomized clinical trial will be conducted in partnership with 2 nursing home corporations who operate a combined total of 142 diverse urban and rural facilities in 8 states. The aims of the 42 month R33 phase are to: 3) Evaluate the primary outcome of hospital transfers over 12 months among patients with dementia in intervention versus control nursing homes; and 4) Compare measures of quality of care at the end of life between the intervention versus control nursing homes. If successful, the APPROACHES ACP Specialist Program will be primed for rapid translation into nursing home practice to reduce unwanted, burdensome hospitalizations and improve quality of care for patients with dementia. Actual enrollment and outcomes will not be available until Centers for Medicare & Medicaid Services (CMS) claims and Minimum Data Set (MDS) data become available. Actual trial enrollment numbers will be updated at that time.

ELIGIBILITY:
Inclusion Criteria:

* Facilities are owned by NH corporate partners
* Facilities are Medicare/Medicaid-certified
* Facilities have an electronic medical records system
* Minimum bedsize of 50 or more;
* At least 50% long-stay as defined by a length of stay of 100 days or longer.

Exclusion Criteria:

* Problematic or unstable facilities will be removed in consultation with NH corporate leaders prior to randomization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47396 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2022-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan Hickman, PhD, Principal Investigator — Indiana University
Locations (2):
- United States (2):
  - Miller's Merry Manor, Warsaw, Indiana
  - Signature HealthCARE LLC, Louisville, Kentucky

REFERENCES:
- [Derived] Hickman SE, Mitchell SL, Hanson LC, Tu W, Stump TE, Unroe KT. The design and conduct of a pragmatic cluster randomized trial of an advance care planning program for nursing home residents with dementia. Clin Trials. 2022 Dec;19(6):623-635. doi: 10.1177/17407745221108992. Epub 2022 Jul 10. PMID 35815777

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 145 nursing homes (NH) in 10 states were screened for eligibility. 142 nursing home (NH) facilities in 8 states met inclusion criteria and were randomized to two arms of the study. Corporate ownership divested from 14 facilities prior to study implementation and were thus excluded from study participation. 128 NHs participated in study implementation and were analyzed.
Pre-assignment Details: The analysis sample is residents who were identified to have Alzheimer's disease or related dementia (ADRD) or a Cognitive Function Scale (CFS) score >=2 and this sample had to be identified after the intervention period through cleaning the resident data received from Centers for Medicare and Medicaid Services (CMS). This is why we had available information for all residents (47396) but only analyzed the sample of ADRD residents (14832). Participant Flow is used to show steps of exclusion.
Units Other Than Participants: Nursing Home Facilities
Period: Overall Study
Arm/Group | APPROACHES ACP Specialist Program | Control
Started (All residents who were living in randomized nursing homes during the study period.) | 24148; 64 Nursing Home Facilities | 23248; 64 Nursing Home Facilities
Completed | 7474; 64 Nursing Home Facilities | 7358; 64 Nursing Home Facilities
Not Completed | 16674; 0 Nursing Home Facilities | 15890; 0 Nursing Home Facilities
Not completed — Resident could not be linked to CMS data | 594 | 435
Not completed — Resident cognitive status could not be determined from CMS data | 6551 | 6426
Not completed — Resident was enrolled in hospice care at study start (exclusion criteria) | 247 | 260
Not completed — Resident did not reside in facility for at least one day of study period (exclusion criteria) | 896 | 573
Not completed — Resident did not have ADRD as defined by study (exclusion criteria) | 8386 | 8196

BASELINE CHARACTERISTICS:
Population: There were 31414 residents residing in participating nursing homes (NH), 15860 in APPROACHES ACP Specialist Program and 15554 in Control. The subpopulation of interest for analysis is residents identified to have Alzheimer's disease, dementia or a Cognitive Function Scale (CFS) score of >=2, therefore the population reported is 7474 residents in APPROACHES ACP Specialist Program and 7358 in Control for a total of 14832.
Groups:
- Total: Total of all reporting groups
Arm/Group | APPROACHES ACP Specialist Program | Control | Total
Number analyzed (Participants) | 7474 | 7358 | 14832
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 759 | 681 | 1440
  >=65 years | 6715 | 6677 | 13392
Age, Continuous [Mean (Standard Deviation); unit: years] | 78.7 (11) | 79.3 (10.8) | 79.0 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4688 | 4683 | 9371
  Male | 2786 | 2675 | 5461
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 318 | 167 | 485
  Not Hispanic or Latino | 7156 | 7191 | 14347
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 3 | 5
  Asian | 6 | 12 | 18
  Native Hawaiian or Other Pacific Islander | 2 | 0 | 2
  Black or African American | 933 | 824 | 1757
  White | 5650 | 5751 | 11401
  More than one race | 13 | 21 | 34
  Unknown or Not Reported | 868 | 747 | 1615
Region of Enrollment [Number; unit: participants]
  United States | 7474 | 7358 | 14832

OUTCOME MEASURES:

1. Primary Outcome: Hospital Transfers
Description: Hospital transfers (admissions and emergency department visits) over 12 months between Alzheimer's Disease and Related Dementias (ADRD) patients in intervention vs. control NHs
Time Frame: 12 months
Population: Only the residents who were identified by our definition as being diagnosed with ADRD are included in our outcomes analyses.
Measure: Mean (Standard Deviation); unit: number of hospital transfers
Arm/Group | APPROACHES ACP Specialist Program | Control
Number analyzed (Participants) | 7474 | 7358
number of hospital transfers | 1.2 (2.3) | 1.3 (2.4)
Statistical Analysis 1: Comparison: APPROACHES ACP Specialist Program vs Control; Test type: Superiority; p = 0.3313, Poisson Regression; Incidence Rate Ratio (IRR) = 0.94, 95% CI 2-sided [0.84 to 1.06], Standard Error of Mean 0.061

2. Secondary Outcome: Hospice Enrollment
Description: % ADRD patients who use hospice
Time Frame: 12 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | APPROACHES ACP Specialist Program | Control
Number analyzed (Participants) | 7474 | 7358
Participants | 1095 | 1181
Statistical Analysis 1: Comparison: APPROACHES ACP Specialist Program vs Control; Test type: Superiority; p = 0.3327, Regression, Logistic; Odds Ratio (OR) = 0.92, 95% CI 2-sided [0.78 to 1.09]

3. Secondary Outcome: Death in Hospital
Description: % ADRD decedents who died in the hospital
Time Frame: 12 months
Population: Only the residents who were identified by our definition as being diagnosed with ADRD are included in our outcomes analyses. Numbers are reported only for participants whose location of death could be confirmed. Participants analyzed is ADRD deaths.
Measure: Count of Participants; unit: Participants
Arm/Group | APPROACHES ACP Specialist Program | Control
Number analyzed (Participants) | 2,005 | 1,980
Participants | 163 | 146
Statistical Analysis 1: Comparison: APPROACHES ACP Specialist Program vs Control; Test type: Superiority; p = 0.3946, Regression, Logistic; Odds Ratio (OR) = 1.13, 95% CI 2-sided [0.85 to 1.49]

ADVERSE EVENTS:
Time Frame: One year
Description: We do not believe that death should be considered an SAE for this trial as: 1) death is often not unexpected in this nursing home population with ADRD; 2) death is not an adverse outcome for patients and families with goals of comfort or palliation if those goals are met; and 3) it is not known whether or not aggressive care provided at the hospital results in lower mortality compared with conservative care in the nursing home
Arm/Group | APPROACHES ACP Specialist Program | Control
All-Cause Mortality (participants affected / at risk) | 2005/7474 | 1980/7358
Serious Adverse Events (participants affected / at risk) | 0/7474 | 0/7358
Other Adverse Events (participants affected / at risk) | 0/7474 | 0/7358

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-07-15): https://cdn.clinicaltrials.gov/large-docs/02/NCT03323502/Prot_SAP_000.pdf